CLINICAL TRIAL: NCT06094231
Title: Treating Patients With Renal Impairment and Altered Glucose MetAbolism With TherapeutIc Carbohydrate Restriction and Sglt2-Inhibiton - a Pilot Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Department of Nephrology Clinic Ottakring Vienna (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRAGMATICS-Pilot
Record Dates: First submitted 2023-10-06; First posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Chronic Kidney Diseases; Diabetes Mellitus; PreDiabetes; Overweight and Obesity
Keywords: Low Carbohydrate Diet; Carbohydrate Restriction; SGLT-2-Inhibitors
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus; Prediabetic State; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional Arm (Experimental): The patients randomized to the interventional Arm will be simultaneously treated with therapeutic carbohydrate restriction and dapagliflozin for a period of three months. During this time repeated measurements of blood ketone levels and a continuous glucose monitoring will be performed.
  Interventions: Behavioral: Therapeutic carbohydrate restriction combined with an SGLT-2-Inhibitor
- Control Arm (No Intervention): The patients randomized to the control arm will continue to receive the standard of care for chronic kidney disease and prediabetes or diabetes, which includes the use of dapagliflozin.

INTERVENTIONS:
Behavioral: Therapeutic carbohydrate restriction combined with an SGLT-2-Inhibitor — The patients will be educated on how to implement a therapeutic carbohydrate restriction, which consists of 50 to 130 grams of carbohydrate per day, simultaneously they will continue to receive the SGLT-2-Inhibitor dapagliflozin.
  Arms: Interventional Arm

SUMMARY:
This randomized controlled trail will evaluate the efficacy and safety of a simultaneous therapeutic carbohydrate restriction and treatment with the Sodium-Glucose-Transporter-2-Inhibitor dapagliflozin in comparison to the standard of care treatment in patients with chronic kidney disease and prediabetes or type 2 diabetes mellitus.

Participants will be randomized 1:1. The interventional group will be educated on how to implement a therapeutic carbohydrate restriction (50-100 grams of carbohydrates per day). Regarding safety, the patients of the interventional group will be provided with continuous glucose monitoring systems and blood ketone meters. The participants of the control group will continue to receive the standard of care therapy for the treatment of chronic kidney disease and prediabetes or type 2 diabetes mellitus. Both groups will be treated with dapagliflozin.

ELIGIBILITY:
Inclusion Criteria:

* Chronic Kidney Disease Stage KDIGO 3a-4 (eGFR eGFR 25-59 mg/min/1.73m²)
* Prediabetes or Diabetes according to the Guideline of the American Diabetes Association (HbA1c >5,7 percent, or fasting glucose values > 100 mg/dL, or glucose levels > 140 mg/dL at 2h during an oral glucose tolerance test)
* Being overweight (Body Mass Index > 25.0 kg/m²)
* Being able to independently:
* - Perform measurements of blood glucose and ketone levels
* - Use a continous glucose monitor
* - Contact the study team

Exclusion Criteria:

* Patients who are allergic to SGLT-2-Inhibitors
* Patients with autoimmune diabetes (Typ 1 or LADA)
* Patients with pancreoprivic diabetes
* Patients with a history of ketoacidosis or lactate acidosis
* Patients with severe hypoglycemic episodes in the 6 moths prior to inclusion
* Patients with bariatric surgery (in the past or planed)
* Patients with nephritic range proteinuria (>3,5g of Albumin/day)
* Patients with active malignant diseases
* Pregnant or breastfeeding patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-25 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Changes in HbA1c | after 3 Months
  Primary endpoint is difference in HbA1c after 3 months in the interventional group

SECONDARY OUTCOMES:
Body composition | after 3 Months
  Body composition will be measured with a body composition monitoring device before and after the study period
Body weight | after 3 Months
  Body weight will be measured before and after the study period
Serum creatinine | after 3 Months
  Serum creatinine will be measured before and after the study period
Serum Cystatin C | after 3 Months
  Serum Cystatin C will be measured before and after the study period
Albuminuria | after 3 Months
  Albuminuria will be measured before and after the study period
Oral glucose tolerance | after 3 Months
  Oral glucose tolerance will be assessed using a 75g oral glucose tolerance test before and after the study period
Glucose variability | during the 3 Months of the study period
  Glucose variability will be assessed using continuous glucose monitor
Time in range | during the 3 Months of the study period
  Time in range regarding glucose will be assessed using continuous glucose monitor

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Scherr, MD, Principal Investigator — 6th Medical Department with Nephrology and Dialysis, Clinik Ottakring, Vienna, Austria
Locations (1):
- 6th Medical Department with Nephrology and Dialysis, Clinik Ottakring, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided